CLINICAL TRIAL: NCT05354037
Title: Flapless Approach for the Treatment of Self-contained Intrabony Defects: a Randomized Controlled Clinical Trial
Brief Title: Flapless Approach for the Treatment of Intrabony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLPERIO
Record Dates: First submitted 2021-09-29; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): EMD + M-MIST approach
  Interventions: Procedure: Enamel matrix derivative application for treatment of intrabony defects
- Group B (Experimental): EMD with flapless approach
  Interventions: Procedure: Enamel matrix derivative application for treatment of intrabony defects

INTERVENTIONS:
Procedure: Enamel matrix derivative application for treatment of intrabony defects — EMD application will be associated to M-MIST approach in control group and flapless approach in test group.

SUMMARY:
The use of Enamel Matrix Derivative (EMD) associated to microsurgical flaps was demonstrated to be effective for the treatment of intrabony defects, in particular in presence of a self-contained anatomy. The main aim of this study will be to evaluate the difference in Clinical Attachment Level (CAL) between baseline and 1-year follow-up, comparing flapless periodontal regeneration using EMD versus the use of EMD after microsurgical flap elevation (Modified-Minimally Invasive Surgical Technique (M-MIST) / Single-flap approach).

DETAILED DESCRIPTION:
The secondary aims of the study are:

* to evaluate the comparative effectiveness of the proposed treatment evaluating patient-centered outcomes.
* to evaluate, after one year from the treatment, the comparative effectiveness evaluating clinical parameters: (I) Probing Depth (PD) measured from the gingival margin to the base of the pocket; (II) Recession (REC) measured as the distance between the CEJ and the gingival margin; (III) Presence of plaque in the site of intervention, measured dichotomously (Yes / No) (Plaque index (PI)); (IV) Presence of bleeding in the site of intervention, measured dichotomously (Yes / No) (Bleeding Index (BI)); (V) Full-mouth Bleeding Score (FMBS%); (VI) Full-mouth Plaque Score (FMPS%); (VII) the proportion of treated sites for each group that presented PD <= 3 mm. ; (VIII) tooth retention
* to evaluate the comparative effectiveness evaluating radiographic parameters: (I) The distance between the Cemento-Enamel Junction (CEJ) and the bottom of the defect (CEJ-A) (II) the distance between the projection of the bone crest to the root surface and the bottom of the defect (representing the intrabony portion of the defect (III) C-A), and the distance between the bone crest and the root surface (representing the maximum width of the defect, C-B) were measured.

Control group: A buccal flap extending to the surfaces of the adjacent teeth will be elevated leading the interdental papilla in position following the M-MIST approach. After degranulation of the defect EMD will be applied following the standard procedure (after preparing root surface with Ethylenediamine tetraacetic acid (EDTA) 22% for two minutes). Non-resorbable 6/0 sutures will be used. The whole procedure will be performed using magnification devices (surgical loupes or surgical microscope). The operator will give postoperative instructions and information about medication.

Test group: The debridement of the pocket will be performed without the elevation of the flap, using ultrasonic tips, air polishing devices and curettes as standard procedure. After that, EMD will be applied and the same procedures as control group will be carried out. Non-resorbable 6/0 sutures will be used in the site of surgical intervention to close coronally the pocket.

At 7 days, suture removal, collection of questionnaires and clinical evaluation will be performed.

Follow-up visits will be carried out at 3, 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over or equal to the age of 18 years
* Patients who are able to understand the requirements of the study and are willing and able to comply with its instructions and schedules
* Patients who had provided written informed consent to participate in the study prior to any study procedure
* Patients in general good health in the opinion of the principal investigator as determined by medical history and clinical examination (American Society of Anesthesiologists ASA 1 or ASA-2)
* Patients having one or more self-contained (3-wall or 2-3 walls) intrabony periodontal defect with an intrabony component of equal or more than 3 mm, as diagnosed by periapical radiographs and clinical evaluation.

Exclusion Criteria:

* FMPS% > 15%
* FMBS% > 15%
* Treatment with anticoagulant drugs (International Normalized Ratio (INR) above 2,5)
* Treatment with intravenous bisphosphonates
* Treatment with anticonvulsants drugs
* untreated Periodontal disease and inability of the patient to maintain reasonable oral hygiene according to study requirements
* Patients with history of alcohol, narcotics or drug abuse
* Patients receiving radiotherapy, chemotherapy or any other immunosuppressive treatment or who have been administered radiotherapy in the last 5 years
* Patients through at any time received radiotherapy to the head and neck region will be excluded anyway
* Uncontrolled bleeding disorders such as: hemophilia, thrombocytopenia, granulocytopenia
* Degenerative diseases
* Osteoradionecrosis
* Renal failure
* Organ transplant recipients
* HIV positive (self-declaration)
* Malignant diseases
* Diseases that compromise the immune system
* Unbalanced diabetes (HbA1c above 7.2 assessed by self-declaration)
* Psychotic diseases
* Hypersensitivity or specific contraindications to one of the components of EMD
* Women who are pregnant (self-declaration); or lactating at the time of recruitment and of surgery
* Site where a history of failed periodontal regenerative procedure in the last two years
* Heavy Smokers (10 cigarettes and more per day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Difference in CAL between baseline and 1-year follow-up | 1 year
  The difference between CAL values at baseline and after 1 year; CAL is defined as the distance between CEJ and the most apical extent of the pocket / sulcus

SECONDARY OUTCOMES:
Difference in PD between baseline and 1-year follow-up | 1 year
  The difference between PD values at baseline and after 1 year; PD is defined as the distance between the gingival margin and the most apical extent of the pocket / sulcus
Difference in REC between baseline and 1-year follow-up | 1 year
  The difference between REC values at baseline and after 1 year; REC is defined as the distance between the CEJ and the gingival margin
Difference in PI between baseline and 1-year follow-up | 1 year
  The difference between PI values at baseline and after 1 year; PI value is 1 if we can detect the presence of plaque or 0 if not
Difference in BI between baseline and 1-year follow-up | 1 year
  The difference between BI values at baseline and after 1 year; BI value is 1 if we can detect the presence of bleeding or 0 if not
Difference in FMBS% between baseline and 1-year follow-up | 1 year
  The difference between FMBS% values at baseline and after 1 year; FMBS% is calculated as the percentage of sites in the whole mouth presenting bleeding
Difference in FMPS% between baseline and 1-year follow-up | 1 year
  The difference between FMPS% values at baseline and after 1 year; FMPS% is calculated as the percentage of sites in the whole mouth presenting plaque
Proportion of treated sites for each group that presented PD <= 3 mm | 1 year
  The number of sites in the whole mouth with PD equal or less than 3 mm
Tooth retention | 1 year
  The presence of tooth in position without any sign / symptom of acute inflammation (abscess, periodical periodontitis)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Corbella, Principal Investigator — University of Milan
Locations (1):
- Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided